CLINICAL TRIAL: NCT05361642
Title: Comparison Between Combined Regional Nasal Block and General Anesthesia Versus General Anesthesia With Dexmedetomidine During Endoscopic Sinus Surgery
Brief Title: Regional Nasal Block and Dexmedetomidine in Endoscopic Sinus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FMASU MD 60/2021
Record Dates: First submitted 2022-02-05; First posted 2022-05-05 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Drug Use
MeSH Terms: interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- regional nasal block (Active Comparator): sphenopalatine ganglion block with general anesthesia
  Interventions: Drug: Bupivacaine HCl 0.5% Injectable Solution
- dexmedetomidine (Active Comparator): use the drug with general anesthesia
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine HCl 0.5% Injectable Solution — using nasal block including sphenopalatine ganglion block with general anesthesia to optimize surgical field
  Other Names: Lidocaine 2%
  Arms: regional nasal block
Drug: Dexmedetomidine — using dexmedetomidine with induction of general anesthesia to optimize surgical field
  Arms: dexmedetomidine

SUMMARY:
The purpose is to compare the efficacy of combined regional nasal block and general anesthesia versus general anesthesia with dexmedetomidine during endoscopic sinus surgery in optimizing intraoperative surgical field.

DETAILED DESCRIPTION:
This study will be done to compare between two different techniques including regional nasal block and dexmedetomidine in optimizing intraoperative surgical field according to average category scale

ELIGIBILITY:
Inclusion Criteria:

* Patients of ASA I or ASA II physical status.
* Patients with age 18-65 years.

Exclusion Criteria:

* Patients with physical status ASA III, IV.
* Known allergic reactions to local anesthetics.
* Patients with history for cerebrovascular or coronary insufficiency.
* Patients with infection at the block site.
* Patients with coagulopathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-11-05 (Estimated); Study Completion 2022-12-05 (Estimated)

PRIMARY OUTCOMES:
Optimizing intraoperative surgical field | Up to 6 months
  Comparison between efficacy of the two techniques in optimizing intraoperative surgical field which will be measured using the average category scale(where grade 0 is defined as no bleeding and grade 5 is defined as severe bleeding, constant suctioning required).

SECONDARY OUTCOMES:
Heart rate in beat per minute | Up to 8 months
  The heart rate will be measured in (beat/minute) at the commencement of surgery and at each assessment of the surgical field. The average mean values during the surgical procedures will be calculated in each group.
Blood loss in millilitres | Up to 8 months
  Blood loss will be measured in millilitres as that collected in the suction apparatus and by weight of the nasal swabs.
endtidal sevoflurane concentration in MAC% | Up to 8 months
  Endtidal sevoflurane concentration will be used as an indicator of inhaled anaesthetic dose. Mean end-tidal sevoflurane concentration will be calculated for each patient as the average of all concentrations recorded will be measured in MAC%
phentolamine requirements in milligrams | Up to 8 months
  The total dose of additional hypotensive agent (phentolamine) requirements will be measured in milligrams
Duration of anesthesia in minutes | Up to 8 months
  Duration of anesthesia will be measured in minutes
Pain assessment with visual analogue scale(VAS) | Up to 8 months
  Pain intensity will be measured with a 10-cm visual analogue scale (where 0 is defined as no pain at all and 10 as the worst possible pain) at 2, 6 and 12 hours postoperatively.
Mean blood pressure in mmHg | Up to 8 months
  The mean blood pressure will be measured in mmHg at the commencement of surgery and at each assessment of the surgical field. The average mean values during the surgical procedures will be calculated in each group.
Duration of surgery in minutes | Up to 8 months
  Duration of surgery will be measured in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Nahed Effat Yossef Salama, Professor, Study Chair — Ain Shams University
Locations (1):
- Moustafa Rakha, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
comparison between the two techniques in optimizing surgical field
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: all collected IPD
URL: http://scopus.com